CLINICAL TRIAL: NCT01518647
Title: Treatment of Multi-organ Bodily Distress Syndrome. A Randomized Controlled Trial of the Effects of Acceptance and Commitment Therapy Given as Group Therapy or Workshop Compared to Standard Treatment (Stress-4)
Brief Title: Acceptance and Commitment Therapy for Patients With Multi-organ Bodily Distress Syndrome (Stress-4)
Acronym: Stress-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110265
Record Dates: First submitted 2012-01-13; First posted 2012-01-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Somatisation Disorder; Somatoform Disorders
Keywords: Bodily Distress Syndrome; Medically unexplained symptoms; Functional somatic symptoms; Functional somatic syndromes; Treatment; Acceptance and Commitment Therapy
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Therapy (Experimental): ACT given as conventional group therapy in groups of 7-8 patients 3,5 hours each session, 9 sessions during 3 month
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Workshop (Experimental): ACT given as a one-day workshop with 15 patients with a following individual consultation
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Standard treatment (Active Comparator): Standard treatment is one single advisory consultation given 2 weeks after randomization
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy is a new third wawe cognitive therapy with the key treatment elements: acceptance, personal values and goals

SUMMARY:
The aim of this study is to test the effect of Acceptance and Commitment Therapy (ACT) in patients with long lasting health problems with no known medical explanation, defined as multi-organ Bodily distress syndrome (BDS). ACT treatment is given as two different types of treatment, a 9-session group therapy and a 1-day workshop followed by an individual consultation, and both are compared to standard treatment, which is one single advisory consultation. The study includes 180 patients.

DETAILED DESCRIPTION:
The aim of this study is to test the effect of Acceptance and Commitment Therapy (ACT) in patients with multi-organ Bodily distress syndrome (BDS). BDS is a unifying diagnosis that encompasses a group of closely related conditions such as somatization disorder, fibromyalgia, irritable bowel syndrome and chronic fatigue syndrome. The project consists of a three-armed randomized controlled trial of ACT treatment given as a supplement to standard treatment as either 9-session group therapy or as a 1-day workshop followed by an individual consultation, compared to standard treatment, which is one single advisory consultation.

Primary outcome is patient-rated improvement measured by Clinical Global Improvement Scale (CGI-I). Secondary outcome is functional level (physical, mental and social) measured by the SF-36 Physical Component Summary (PCS). The study includes 180 participants.

ELIGIBILITY:
Inclusion Criteria:

1. First time refered patients fulfilling diagnostic criteria for BDS multi-organ type with symptoms for more than 3 of 4 symptom categories
2. Moderate or severe impact on daily life
3. Symptoms lasting for at least 2 years
4. Age 20-50 years
5. Born in Denmark or have Danish parents. The patient understands, speaks, writes and read Danish.

Exclusion Criteria:

1. Presence og other physical of psychiatric condition, if the symptoms of this condition can not clearly be separated from symptoms of BDS
2. Patients with treatment demanding psychiatric disease as dominating problem
3. A lifetime-diagnosis of psychoses, mania or depression with psychotic symptoms (ICD-10: F20-29, F30-31, F32.3, F33.3)
4. Abuse of alcohol, narcotics or drugs
5. Pregnancy at time of inclusion

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2015-08-25 (Actual); Study Completion 2016-02-09 (Actual)

PRIMARY OUTCOMES:
Global Clinical Improvement Scale | 14 month after randomization
  Questionnaire, patient-rated improvement of health since the beginning of the study.

SECONDARY OUTCOMES:
SF-36 | Before randomization, and at 6, 14 and 20 months after randomization
  Questionnaire, patient-rated. Assessment of physical, social and mental functioning
Visual Analogue Scale for pain and worst symptom | Before randomization, and at 6, 14 and 20 month after randomization
Symptom Checklist (SCL) | Before randomization, and at 6, 14 and 20 month after randomization
  Questionnaire, patient-rated. Assessment of physical, social and mental functioning
WHODAS II | Before randomization, and at 6, 14 and 20 month after randomization
  Questionnaire, patient-rated. Assessment of physical, social and mental functioning

CONTACTS AND LOCATIONS:
Overall Officials: Johanne L Agger, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Research Clinic for Functional Disorders, Aarhus, Denmark